CLINICAL TRIAL: NCT00001396
Title: Obstructive Hypertrophic Cardiomyopathy (HCM) in Children: Natural History and Results of Dual Chamber (DDD) Pacemaker Therapy
Brief Title: Natural History and Results of Dual Chamber (DDD) Pacemaker Therapy of Children With Obstructive Hypertrophic Cardiomyop...
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 940001; 94-H-0001
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-07-23

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: Pacemaker; Pediatric; Obstructive HCM
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

INTERVENTIONS:
Device: Paragon Pacemaker

SUMMARY:
Several studies have shown that specialized pacemaking devices (DDD pacing) can improve the symptoms associated with hypertrophic cardiomyopathy (HCM) in adults. In addition, studies have also shown that specialized pacemaking devices (DDD pacing) can improve conditions of HCM in children. However, growth of the body and organs, including the heart, is very rapid during childhood. Therefore the long-term effects of DDD pacing in children are unknown.

The purpose of this study is to examine the growth rate and nutrition of children with HCM. Due to this heart condition and the restrictions that are often placed on the child's activity level, children with HCM may grow at a slower rat and may have a greater tendency to be overweight.

Children participating in the study will have their growth rate and nutritional status measured before the study begins and throughout the course of the study.

Findings in this research study will not directly benefit the patients participating in it. However, information gathered as a result of this study may lead to improvements in the management of children with HCM in the future.

DETAILED DESCRIPTION:
Several studies have shown that dual chamber (DDD) pacemaker therapy relieves LV outflow obstruction and improves symptoms in most adult patients with obstructive hypertrophic cardiomyopathy (HCM). It is however, uncertain whether DDD pacing will be efficacious in children with obstructive HCM, because of evolving cardiac morphology and increased LV hypertrophy and outflow obstruction associated with rapid body growth. We propose to monitor clinical progress, and cardiac morphologic and hemodynamic changes over several years following implantation of a DDD pacemaker in children who present with obstructive HCM between the ages of 5 to 15 years. Functional status, myocardial ischemia, arrhythmias, and LV outflow obstruction will be evaluated by exercise tests, echocardiography, thallium scintigraphy, Holter monitoring, electrophysiologic and cardiac catheterization studies. The results of pacemaker therapy will be compared with the findings in a cohort of young patients with obstructive HCM who elect not to be treated with DDD pacemaker.

ELIGIBILITY:
* INCLUSION CRITERIA: DDD Pacemaker Therapy

Children of either gender, aged 5 to 15 years.

Presence of LV hypertrophy and LV outflow obstruction.

EXCLUSION CRITERIA: DDD Pacemaker Therapy

Other systemic disease that prevent evaluation by echocardiography or cardiac catheterization.

Chronic atrial fibrillation.

Positive pregnancy test.

INCLUSION CRITERIA: Cohort Study

Children of either gender, 5 to 20 years (children greater than 15 years will be included if there is access to reliable previous catheterization data).

Presence of LV hypertrophy and LV obstruction.

EXCLUSION CRITERIA: Cohort Study

Other systemic disease that prevent evaluation by echocardiography or cardiac catheterization.

Chronic atrial fibrillation.

Positive pregnancy test.

Ages: 5 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100
Dates: Start 1993-10-06; Study Completion 2008-07-23

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Fananapazir L, Cannon RO 3rd, Tripodi D, Panza JA. Impact of dual-chamber permanent pacing in patients with obstructive hypertrophic cardiomyopathy with symptoms refractory to verapamil and beta-adrenergic blocker therapy. Circulation. 1992 Jun;85(6):2149-61. doi: 10.1161/01.cir.85.6.2149. PMID 1350522
- [Background] Slade AK, Sadoul N, Shapiro L, Chojnowska L, Simon JP, Saumarez RC, Dodinot B, Camm AJ, McKenna WJ, Aliot E. DDD pacing in hypertrophic cardiomyopathy: a multicentre clinical experience. Heart. 1996 Jan;75(1):44-9. doi: 10.1136/hrt.75.1.44. PMID 8624871
- [Background] McAreavey D, Fananapazir L. Altered cardiac hemodynamic and electrical state in normal sinus rhythm after chronic dual-chamber pacing for relief of left ventricular outflow obstruction in hypertrophic cardiomyopathy. Am J Cardiol. 1992 Sep 1;70(6):651-6. doi: 10.1016/0002-9149(92)90207-f. PMID 1510015